CLINICAL TRIAL: NCT00423111
Title: Correlation Between Cognitive Functions and MRI in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4487-AA-CTIL
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Memory; Cognitive deficits; MRI; Hippocampus; Prefrontal cortex
MeSH Terms: conditions — Multiple Sclerosis; Cognition Disorders

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The purpose of this study is to determine whether there is a correlation between cognitive functions and volume of specific brain area measured in MRI of multiple sclerosis patients.

DETAILED DESCRIPTION:
Recent literature suggests that multiple sclerosis is accompanied by significant deficits in cognitive performance. The origin of these cognitive deficits is not known, since the severity of cognitive deficits was not found to be correlated with disease parameters such as duration, lesion load or disease intensity as measured on standard scales (e.g. EDSS). The research hypothesis we plan to test is that the individual intensity of cognitive deficits is correlated with degeneration of specific neuronal structures related to cognitive performance, such as the hippocampus and prefrontal cortex.

To test this hypothesis, we plan to perform volumetric measurements of such regions on MRI scans obtained from MS patients during the course of their clinical evaluation, and attempt to correlate those with the results of neuropsychological tests performed by the same subjects around the time of MRI scanning.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Multiple Sclerosis
* Age 18-65

Exclusion Criteria:

* Another brain disease
* Stroke
* Brain trauma
* Neurosurgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-02; Study Completion 2009-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anat Achiron, MD Ph.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel